CLINICAL TRIAL: NCT02666196
Title: A Single Dose-Escalation Study to Evaluate the Safety and Pharmacokinetics of Orally Administered DAA-I in Healthy Subjects
Acronym: DAA-I
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Principal Investigator, Medicine, Professor Lee Kok Onn, Senior Consultant, National University Hospital, Singapore
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: DAA-I
Record Dates: First submitted 2015-12-14; First posted 2016-01-28 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- DAA-I 6mg (Experimental): Subjects given solid compound in vials containing 6mg per vial
  Interventions: Drug: DAA-I
- DAA-I 50mg (Experimental): Subjects given solid compound in vials containing 50mg per vial
  Interventions: Drug: DAA-I
- DAA-I 110mg (Experimental): Subjects given solid compound in vials containing 110mg per vial
  Interventions: Drug: DAA-I
- Placebo (Placebo Comparator): Subjects given 25ml placebo dissolved in 200ml water
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DAA-I
  Arms: DAA-I 110mg; DAA-I 50mg; DAA-I 6mg
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a placebo-controlled randomized phase 1 study to investigate the safety and pharmacokinetics of DAA-I in a cohort of healthy subjects.

DETAILED DESCRIPTION:
The study will be a single-blind, step-wise dose escalation, placebo controlled study in healthy subjects consisting of up to 3 dose steps of DAA-I. In the sequential step wise design, a single dose of DAA-I or placebo will be administered to 6 subjects for one treatment group. For each dose step, 4 subjects will receive DAA-I and 2 subjects will receive placebo. Subjects will be randomly allocated to one dose step. Step One would have to be completed before Step Two. Escalation up to Step Two and subsequent steps would depend on the safety results from the preceding step(s). There will be an interval of 6 hours between the dosing of the first and second DAA-I-treated volunteers of each cohort to allow for early cardiovascular monitoring. Only if there are no safety signals identify from these subjects as assessed by the Safety Review Committee can simultaneous dosing of the remaining volunteers be carried out.

ELIGIBILITY:
Inclusion Criteria:

1. Overtly healthy males or females as determined by medical history and physical examination.
2. Between the ages of 21 and 50 years, inclusive.
3. Weight limits within range of Body Mass Index (BMI) 19-30kg/m2
4. Renal, hepatic and blood chemistry results within normal range.
5. Normal blood pressure and heart rate as determined by the investigator.(Normal range: Systolic BP 100-140mmHg;Diastolic BP 40-90mmHg; Heart rate 50 - 100 beats per minute)
6. Temperature between 36oC to 37.4oC
7. Electrocardiogram considered as within normal limits by the investigator.
8. Are reliable and willing to make themselves available for the duration of the study.
9. Ability to provide informed consent.

Exclusion Criteria:

1. History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, neurological disorders capable of altering the absorption, metabolism or elimination of drugs, or of constituting a risk factor when taking the study medication.
2. Evidence of significant active haematologic disease and/or blood donation in the last 3 months.
3. Are pregnant or intend to become pregnant during the course of the study.
4. Sexually active women of childbearing age not actively practising birth control by using oral contraceptives or an intrauterine device (IUD).
5. Women who are lactating.
6. History of allergic reactions to angiotensin inhibitor (AI), angiotensin II inhibitors, DAA-I or other relevant allergic reactions of any origins.
7. Participation in a study involving administration of an investigational compound within the past 30 days.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2015-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety and dose range of DAA-I after single oral dose administration | 24 hours
  Evaluate the safety (in terms of effect on normal blood pressure, pulse, and 12-lead ECG) of DAA-I following a single oral administration in 12 healthy subjects (0.08 mg/kg/subject in 4 subjects, 0.7 mg/kg/subject in 4 subjects, and 1.5 mg/kg/subject in 4 subjects).

SECONDARY OUTCOMES:
Evaluate the pharmacokinetics of DAA-I after single oral dose administrations | 24 hours
  Evaluate the plasma level of DAA-I in each subject at baseline (0 hr) and at 0.25, 0.5, 1, 2, 3, 4, 5, 6, and 12 hr after oral administration of a single-dose of DAA-I, and determine the area under the plasma concentration versus time curve (AUC).

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee KO, Khoo CM, Chowbay B, Chan YH, Sim MK. A Single Dose-Escalation Study to Evaluate the Safety and Pharmacokinetics of Orally Administered Des-Aspartate Angiotensin I in Healthy Subjects. Drugs R D. 2016 Dec;16(4):317-326. doi: 10.1007/s40268-016-0143-y. PMID 27681888